CLINICAL TRIAL: NCT00729508
Title: A Double-Blind, Randomised, Placebo-Controlled Study to Evaluate the Efficacy of Cat-PAD in Cat Allergic Subjects Following Challenge to Cat Allergen in an Environmental Exposure Chamber.
Brief Title: Effectiveness of Cat-PAD to Treat Cat Allergy in Cat Allergic Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Circassia Limited (Industry)
Responsible Party: Rod Hafner, Circassia Limited
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CP002
Record Dates: First submitted 2008-08-04; First posted 2008-08-07 (Estimated); Last update posted 2009-07-08 (Estimated); Status verified 2009-07

CONDITIONS: Cat Allergy
Keywords: Cat allergy; Immunotherapy; Cat-PAD; Environmental Exposure Chamber

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental)
  Interventions: Biological: Cat-PAD
- 2 (Experimental)
  Interventions: Biological: Cat-PAD
- 3 (Experimental)
  Interventions: Biological: Cat-PAD
- 4 (Experimental)
  Interventions: Biological: Cat-PAD
- 5 (Placebo Comparator)
  Interventions: Biological: Cat-PAD

INTERVENTIONS:
Biological: Cat-PAD — Cat-PAD dose 2X 4 administrations 2 weeks apart
  Arms: 1
Biological: Cat-PAD — Cat-PAD dose 1X 4 administrations 2 weeks apart
  Arms: 2
Biological: Cat-PAD — Cat-PAD dose 1X 4 administrations 4 weeks apart
  Arms: 3
Biological: Cat-PAD — Cat-PAD dose 1X 8 administrations 2 weeks apart
  Arms: 4
Biological: Cat-PAD — Placebo
  Arms: 5

SUMMARY:
Cat allergy is an increasingly prevalent condition, affecting 10-15% of patients with allergic rhinoconjunctivitis and/or asthma. Cat-PAD is a novel, synthetic, allergen-derived peptide desensitising vaccine, currently being developed for the treatment of cat allergy. This study will investigate the efficacy of 4 treatment regimens of Cat-PAD in cat allergic subjects following challenge to cat allergen in an environmental exposure chamber (EEC).

DETAILED DESCRIPTION:
This study is designed as a multicentre, randomised, double-blind, placebo-controlled study of 4 treatment regimens in up to 120 cat allergic subjects. A total of 24 subjects will be randomised into each treatment group. Each subject will undergo screening up to 4 weeks before treatment. Baseline challenge will consist of exposure to cat allergen for 3 hours in an EEC on 4 visits on successive days a week before the first administration of Cat-PAD or placebo. Treatment will be administered as intradermal injections into the flexor surface of alternate forearms. There are 5 treatment regimens involving administration of Cat-PAD or placebo. Post-treatment challenge (PTC) will consist of exposure to cat allergen for 3 hours in an EEC on 4 visits on successive days 18 weeks after the first administration of study medication.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 1-year documented history of rhinoconjunctivitis (Nasal symptoms: sneezing, itching, rhinorrhoea, blockage; Ocular symptoms: itching, redness, soreness, watering) on exposure to cats. [Subjects may also have controlled asthma (GINA classification 1)].
* Positive skin prick test to cat allergen with a wheal diameter at least 3mm larger than that produced by the negative control.
* Subjects must achieve minimum qualifying symptom scores on at least one Symptom Diary Card during EEC exposure on the third and fourth day during the Baseline Challenge. Minimum qualifying symptom scores are defined as a TRSS of at least 10 out of a possible 24 and a TNSS of at least 6 out of a possible 12.

Exclusion Criteria:

* Subjects with asthma falling under GINA classification 2 (partly controlled) and 3 (uncontrolled).
* A history of anaphylaxis to cat allergen.
* Subjects with a cat specific IgE >100 kU/L.
* Subjects with an FEV1 <80% of predicted.
* Subjects with an acute phase skin response to cat allergen with a mean wheal diameter > 50mm.
* Subjects who suffer from seasonal allergic rhinoconjunctivitis, and cannot complete the clinical study outside the local pollen season or who have significant allergy to other animal dander that cannot be avoided during the study period.
* Subjects who cannot tolerate baseline challenge in the EEC.
* Allergen immunotherapy during the last 12 months or any history of Cat Dander immunotherapy.
* Subjects for whom administration of adrenaline is contra-indicated (e.g. subjects with acute or chronic symptomatic coronary heart disease or severe hypertension).
* Subjects being treated with beta-blockers.
* History of immunopathological diseases.
* Positive test for Hepatitis B, Hepatitis C or HIV at screening.
* Have a history of severe drug allergy or anaphylactic reaction to food.
* A known allergy to thioglycerol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2008-08; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in Total Rhinoconjunctivitis Symptom Score (TRSS) using all timepoints during PTC in Cat-PAD treatment groups compared to placebo. | 18 weeks

SECONDARY OUTCOMES:
Change from baseline in TRSS in Cat-PAD treatment groups at last two timepoints on third and fourth challenge days compared to placebo. | 18 weeks
Change from baseline in individual symptom scores for ocular and nasal symptoms at all timepoints during Exposure Chamber visit in Cat-PAD treatment groups compared to placebo. | 18 weeks
Change from baseline in TRSS at all timepoints during Exposure Chamber visit in pooled data from Cat-PAD treatment groups compared to placebo. | 18 weeks
Proportion of subjects prematurely leaving the EEC due to intolerable symptoms during Post-Treatment Challenge (PTC) in Cat-PAD treatment groups compared to placebo. | 18 weeks
Change from baseline in EEC-Rhinoconjunctivitis Quality of Life Questionnaire (EEC-RQOL) at all timepoints during Exposure Chamber visit in Cat-PAD treatment groups compared to placebo. | 18 weeks
Exploratory analyses of change from baseline in asthma symptoms, FEV1 and use of rescue medication in Cat-PAD treatment groups compared to placebo in asthmatic subjects. | 18 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Deepen Patel, MD, Principal Investigator — Allied Research International Inc-Cetero Research
Locations (1):
- Cetero Research, Toronto, Ontario, Canada